CLINICAL TRIAL: NCT00350246
Title: Long-term Effects of Laser Refractive Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 66-04
Record Dates: First submitted 2006-07-07; First posted 2006-07-10 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

INTERVENTIONS:
Procedure: Laser Refractive Surgery

SUMMARY:
This study will determine if there are short- and long-term postoperative differences in visual and corneal outcomes between different laser refractive surgical procedures.

DETAILED DESCRIPTION:
We will measure postoperative differences in visual acuity, contrast sensitivity, corneal light scatter, density of keratocytes and subbasal nerves, corneal sensitivity, corneal topography and wavefront between PRK performed with epithelial removal by a laser or by a rotary brush and between LASIK performed by using a microkeratome or by using a femtosecond laser. Measurements will be made at baseline and at intervals over 5 postoperative years in 21 LASIK patients, 20 PRK patients, and 20 unoperated controls.

ELIGIBILITY:
Myopia 1-10 diopters No other ocular abnormalities except presbyopia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
keratocyte density at 5 years
nerve density at 5 years

CONTACTS AND LOCATIONS:
Overall Officials: William M. Bourne, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Patel SV, McLaren JW, Kittleson KM, Bourne WM. Subbasal nerve density and corneal sensitivity after laser in situ keratomileusis: femtosecond laser vs mechanical microkeratome. Arch Ophthalmol. 2010 Nov;128(11):1413-9. doi: 10.1001/archophthalmol.2010.253. PMID 21060042
- [Derived] Calvo R, McLaren JW, Hodge DO, Bourne WM, Patel SV. Corneal aberrations and visual acuity after laser in situ keratomileusis: femtosecond laser versus mechanical microkeratome. Am J Ophthalmol. 2010 May;149(5):785-93. doi: 10.1016/j.ajo.2009.12.023. Epub 2010 Mar 15. PMID 20227675